CLINICAL TRIAL: NCT04728919
Title: Nasal and Pulmonary Nitric Oxide Output in COVID-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Lauri Lehtimäki, associate professor, Tampere University Hospital
Other Study IDs: R200090
Record Dates: First submitted 2021-01-19; First posted 2021-01-28 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive cases: Subjects with acute respiratory infection and positive COVID-19 test, who are well enough to be treated at home.
- COVID-19 negative controls: Subjects with acute respiratory infection and negative COVID-19 test, who are well enough to be treated at home.

SUMMARY:
A Study of the relation of COVID-19 infection and its severity to upper and lower airway nitric oxide, upper airway viral load and lung function.

DETAILED DESCRIPTION:
Materials and methods: Prospective cohort of 40 COVID-19, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), positive patients from Tampere university hospital region are recruited to the study. Forty COVID-19 negative patients with similar symptoms act as a control group.

All subjects are screened for other respiratory viruses with reverse transcriptase polymerase chain reaction (RT-PCR)-multiplex tests. Viral loads of SARS-CoV-2 from anterior nasal cavity, nasopharynx, throat and saliva are evaluated by RT-PCR cycle treshold (Ct) value and antigen testing (RLU value).

During the first visit NEWS (National Early Warning Score), recorded pulmonary auscultation (Thinklabs One, Thinklabs Medical LLC), impulse oscillometry (Tremoflo, THORASYS Thoracic Medical Systems Inc), FeNO (fractional exhaled nitric oxide) and FnNO (fractional nasal nitric oxide) (NIOX VERO®,Circassia) are conducted. All aforementioned and a spirometry are measured again after 2 months.

Aims: To evaluate the relation of COVID-19 infection and its severity to upper and lower airway nitric oxide, viral load and lung function. To compare the capability of RT-PCR in detecting SARS-CoV-2 RNA from saliva, anterior nasal swab samples and oropharyngeal swap samples vs. the golden standard of nasopharyngeal swab samples. To compare the results of RT-PCR and antigen test in detecting SARS-CoV-2 from nasal and pharyngeal sample sites.

ELIGIBILITY:
Inclusion Criteria:

* capable of breathing through nose, no need of supplemental oxygen, symptom onset within 10 days, positive SARS-CoV-2 test in Fimlab and capable of performing all required tests

Exclusion Criteria:

* need of supplemental oxygen, pregnancy, lactation, incapability of performing the tests for any reason, use of organic nitrate medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms of COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Viral load of SARS-CoV-2 from different sample sites | 0 months
  RT-PCR (Ct value) and antigen testing (RLU value)
Upper respiratory tract viruses | 0 months
  RT-PCR-multiplex tests, from nasopharyngeal sample site
FeNO | Baseline
  Fractional exhaled nitric oxide in ppb obtained NIOX VERO
FnNO | Baseline
  Nasal nitric oxide in ppb obtained NIOX VERO
FeNO | 2 months
  Fractional exhaled nitric oxide in ppb obtained NIOX VERO
Change in FeNO | BAseline and at 2 months
  FeNO at 2 months - FeNO at baseline
FnNO | 2 months
  Nasal nitric oxide in ppb obtained NIOX VERO
CHange in FnNO | Baseline and at 2 months
  FnNO at 2 moths - FnNO at baseline
Airway resistance at 20Hz, R20 | Baseline
  Airway resistance at 20Hz obtained from Impulse oscillometry
Airway resistance at 5Hz, R5 | Baseline
  Airway resistance at 5Hz obtained from Impulse oscillometry
Airway resistance at 20 Hz, R20 | 2 months
  Airway resistance at 20 Hz obtained from Impulse oscillometry
Change in R20 | Baseline and at 2 months
  R20 at 2 months - R20 at baseline
Airway resistance at 5Hz, R5 | 2 months
  Airway resistance at 5Hz obtained from Impulse oscillometry
Change in R5 | Baseline and at 2 months
  R5 at 2 months - R5 at baseline
Reactance at 5Hz (X5) | Baseline
  Airway reactance at 5 Hz obtained from Impulse oscillometry
Reactance at 5Hz (X5) | 2 months
  Airway reactance at 5 Hz obtained from Impulse oscillometry
Change in X5 | Baseline and at 2 months
  X5 at 2 months - X5 at baseline
Resonant frequency (Fres) | Baseline
  Resonant frequency (Fres) obtained from Impulse oscillometry
Resonant frequency (Fres) | 2 months
  Resonant frequency (Fres) obtained from Impulse oscillometry
Change in Fres | Baseline and at 2 months
  Fres at 2 months - Fres at baseline
Reactance area (AХ) | Baseline
  Reactance area (AХ) obtained from Impulse oscillometry
Reactance area (AХ) | 2 months
  Reactance area (AХ) obtained from Impulse oscillometry
Change in AX | Baseline and at 2 months
  AX at 2 months - AX at baseline

SECONDARY OUTCOMES:
FEV1 | 2 months
  Forced expiratory volume in 1 second
FVC | 2 months
  Forced vital capacity
VC | 2 months
  Vital capacity
FEV1/FVC | 2 months
  Forced expiratory volume in 1 second divided by forced vital capacity
FEV1/VC | 2 months
  Forced expiratory volume in 1 second divided by vital capacity

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Lehtimäki, Professor, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland